CLINICAL TRIAL: NCT06731998
Title: Evaluating Optimal Perioperative Pain Management: A Prospective Randomized Control Trial of Laparoscopic Transversus Abdominis Plane Block With Local Anesthetic, Laparoscopic Transversus Abdominis Plane Block Alone, and Local Anesthetic Alone in Minimally Invasive Oncologic Surgery
Brief Title: Optimal Perioperative Pain Control in Minimally Invasive Abdominal Cancer Surgery
Acronym: LapTAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Casey Allen, MD, Assistant Professor, Surgical Oncologist, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LapTAP
Record Dates: First submitted 2024-11-12; First posted 2024-12-13 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Oncologic Surgery; Cancer; Cancer Surgery; Hepatic Cancer; Gastric (Cardia, Body) Cancer; Biliary Tract Cancer; Pancreatic Cancer Resectable; Gynecologic Cancers; Gastrointestinal Cancers; Colorectal Cancer; Minimally Invasive Surgical Procedures
Keywords: Laparoscopic Transversus Abdominis Plane Block; Local Anesthetic; Laparoscopic Surgical Procedure; pain management; cancer; cancer surgery; oncologic surgery; perioperative pain management; minimally invasive surgical procedures
MeSH Terms: conditions — Neoplasms; Liver Neoplasms; Biliary Tract Neoplasms; Gastrointestinal Neoplasms; Colorectal Neoplasms; Agnosia | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Laparoscopic Transversus Abdominis Plane Block with Local Anesthetic (Active Comparator): Patient would be receiving Laparoscopic Transversus Abdominis Plane block in addition to Local Anesthetic per standard of care.
  Interventions: Procedure: Local Anesthesia; Procedure: Laparoscopic Transversus Abdominis Plane block
- Laparoscopic Transversus Abdominis Plane block only (Active Comparator): Patient would be receiving Laparoscopic Transversus Abdominis Plane block without Local Anesthetic per standard of care.
  Interventions: Procedure: Laparoscopic Transversus Abdominis Plane block
- Local Anesthetic only (Active Comparator): Patient would be receiving Local Anesthetic per standard of care.
  Interventions: Procedure: Local Anesthesia

INTERVENTIONS:
Procedure: Local Anesthesia — For local anesthetic administration at port sites, 30 mL of 0.1% ropivacaine is injected around the umbilical port site following the completion of the primary surgical procedure. Additionally, 5 mL of 0.1% ropivacaine is injected around each additional port site to ensure effective local anesthesia.
  Arms: Laparoscopic Transversus Abdominis Plane Block with Local Anesthetic; Local Anesthetic only
Procedure: Laparoscopic Transversus Abdominis Plane block — Surgeon will place 18 gauge needle into the fascial plane between the internal oblique and transversus abdominis muscles. Once the needle is accurately positioned surgeon will inject 15 mL of 0.1% ropivacaine slowly. This procedure is performed bilaterally to ensure comprehensive analgesia. The total volume utilized for the LapTAP block is 30 mL of 0.1% ropivacaine.
  Arms: Laparoscopic Transversus Abdominis Plane Block with Local Anesthetic; Laparoscopic Transversus Abdominis Plane block only

SUMMARY:
This is a research study to evaluate the effectiveness of 3 different types of routine pain management regimens used during clinically indicated, minimally invasive oncologic (cancer) surgery. This project is considered "Research" and participation is voluntary. Upon enrollment in this study, the research team will collect data from the patient's medical records. The patient will undergo all of the normal testing and procedures required pre-operatively (standard of care). The study team will then randomly assign the patient (like a flip of a coin) to one of three different study arms for pain management during surgery:

1. Laparoscopic Transversus Abdominis Plane Block (LapTAP) with Local Anesthetic (LA)
2. Laparoscopic Transversus Abdominis Plane Block (LapTAP) only
3. Local Anesthetic (LA) only The patient will receive standard pre- and post-operative care according to clinical guidelines (routine care). The study team will collect information from the patient's medical record for the first 24 hours after their surgery and upon discharge. This information will include pain scores, amount of medication required, any side effects the patient may have experienced, and satisfaction with pain control. Participation in the study will end upon discharge from the hospital.

DETAILED DESCRIPTION:
Traditional pain management strategies have heavily relied on the use of Local Anesthesia (LA). Laparoscopic Transversus Abdominis Plane block (LapTAP) has emerged as a new approach for postoperative pain control following minimally invasive surgery, promising enhanced pain control in comparison with traditional approaches. Preliminary investigations into LapTAP have shown promise, yet there remains a significant gap in comparative effectiveness research, especially juxtaposed against the more traditional LA. We propose a comprehensive three-arm superiority trial evaluating LapTAP in conjunction with LA, LapTAP alone, and LA alone. We intend to scrutinize the efficacy of each modality in managing postoperative pain specific to minimally invasive oncologic surgery. Findings from this trial will be used to refine clinical protocols, improve patient outcomes, and potentially standardize care in postoperative pain management for minimally invasive oncologic procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age ≥ 18 - 89
2. Patients scheduled for elective (clinically indicated) hepatic, gastric, biliary, pancreatic, gynecologic, colorectal, other GI Minimally invasive oncologic surgery.
3. Patients who have provided informed consent to participate in the study.
4. Patients with an American Society of Anesthesiologists (ASA) physical status classification of I, II, or III.
5. Patients undergoing procedures anticipated to last more than 1 hour but less than 8 hours.
6. Patients able to understand and self-report pain using the designated pain Visual Analog Scale

Exclusion Criteria:

1. Patients age less than 18 or ≥ 90
2. Pre-existing hepatic dysfunction, cirrhosis
3. Patients with an ASA classification of IV or higher.
4. Patients with chronic pain disorders or on long-term opioid or analgesic therapy.
5. Patients with known contraindications to the study drugs or procedures (e.g., allergy to LA or contraindications to LapTAP).
6. Patients with cognitive impairments or psychiatric conditions that could interfere with pain assessment or understanding of informed consent.
7. Patients unable to understand the language in which consent and study-related information are provided (The study and the study-related information will be in the English Language)..
8. Patients who have undergone major surgery within the last 6 months.
9. Female patients who are pregnant.
10. Patients currently enrolled in another clinical trial that might interfere with the outcome measures of this study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain Score | Hourly, starting 1 hour post surgery for 24 hours, then at time of hospital discharge (on average 1 week)
  Pain will be measured in the post anesthesia care unit (PACU) using Visual Analog Scale. Pain will be scored from zero to ten, with zero being no pain at all and ten being unbearable pain.

SECONDARY OUTCOMES:
Opioid Consumption | up to 24 hours post surgery
  Opioid consumption (milligrams) within the first 24 hours post-surgery (standardize with Morphine equivalence).
Recovery Analgesic Time | up to 24 hours post surgery
  Time to first rescue analgesic request
Adverse Event(s) Frequency | immediately post surgery up through discharge (on average of 1 week)
  Frequency of any adverse events related to interventions
Adverse Event(s) Severity | immediately post surgery up through discharge (on average of 1 week)
  Severity of any adverse events related to interventions
Patient Satisfaction with Pain Management | At discharge (on average of 1 week)
  Will gauge patient perceptions of pain control and overall satisfaction with their treatment with a standardized Visual Analog Scale utilizing a zero to ten scale, with zero being completely dissatisfied and ten being completely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Casey Allen, MD, Principal Investigator — Allegheny Health Network
Locations (1):
- AHN West Penn Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
It is not necessary for the scope of the study to share IPD.

REFERENCES:
- [Background] 17. https://pain.ucsf.edu/fascial-plane-blocks/transversus-abdominis-plane-tap-block
- [Background] Jones JH, Aldwinckle R. Interfascial Plane Blocks and Laparoscopic Abdominal Surgery: A Narrative Review. Local Reg Anesth. 2020 Oct 23;13:159-169. doi: 10.2147/LRA.S272694. eCollection 2020. PMID 33122942
- [Background] Guo Q, Li R, Wang L, Zhang D, Ma Y. Transversus abdominis plane block versus local anaesthetic wound infiltration for postoperative analgesia: A systematic review and meta-analysis. Int J Clin Exp Med. 2015 Oct 15;8(10):17343-52. eCollection 2015. PMID 26770326
- [Background] Hamid HK, Emile SH, Saber AA, Ruiz-Tovar J, Minas V, Cataldo TE. Laparoscopic-Guided Transversus Abdominis Plane Block for Postoperative Pain Management in Minimally Invasive Surgery: Systematic Review and Meta-Analysis. J Am Coll Surg. 2020 Sep;231(3):376-386.e15. doi: 10.1016/j.jamcollsurg.2020.05.020. Epub 2020 Jun 2. PMID 32502615
- [Background] Siddiqui MR, Sajid MS, Uncles DR, Cheek L, Baig MK. A meta-analysis on the clinical effectiveness of transversus abdominis plane block. J Clin Anesth. 2011 Feb;23(1):7-14. doi: 10.1016/j.jclinane.2010.05.008. PMID 21296242
- [Background] Mannava S, Hafezi N, Turk F, Colgate C, Askegard-Giesmann J, Markel T, Horn N, Gray B. Transversus Abdominis Plane Block VS. Local Wound Infiltration for Elective Minimally Invasive Cholecystectomy in Children: A Prospective Randomized Trial. J Pediatr Surg. 2024 Jan;59(1):96-102. doi: 10.1016/j.jpedsurg.2023.09.020. Epub 2023 Sep 22. PMID 37863700
- [Background] Calle GA, Lopez CC, Sanchez E, De Los Rios JF, Vasquez EM, Serna E, Arango AM, Castaneda JD, Vasquez RA, Gonzalez A, Escobar A, Almanza LA. Transversus abdominis plane block after ambulatory total laparoscopic hysterectomy: randomized controlled trial. Acta Obstet Gynecol Scand. 2014 Apr;93(4):345-50. doi: 10.1111/aogs.12351. PMID 24575769
- [Background] Rajanbabu A, Puthenveettil N, Appukuttan A, Asok A. Efficacy of laparoscopic-guided transversus abdominis plane block for patients undergoing robotic-assisted gynaecologic surgery: A randomised control trial. Indian J Anaesth. 2019 Oct;63(10):841-846. doi: 10.4103/ija.IJA_471_19. Epub 2019 Oct 10. PMID 31649397
- [Background] El Hachem L, Small E, Chung P, Moshier EL, Friedman K, Fenske SS, Gretz HF 3rd. Randomized controlled double-blind trial of transversus abdominis plane block versus trocar site infiltration in gynecologic laparoscopy. Am J Obstet Gynecol. 2015 Feb;212(2):182.e1-9. doi: 10.1016/j.ajog.2014.07.049. Epub 2014 Aug 1. PMID 25088860
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Ye SP, Zhu WQ, Huang ZX, Liu DN, Wen XQ, Li TY. Role of minimally invasive techniques in gastrointestinal surgery: Current status and future perspectives. World J Gastrointest Surg. 2021 Sep 27;13(9):941-952. doi: 10.4240/wjgs.v13.i9.941. PMID 34621471
- [Background] Small C, Laycock H. Acute postoperative pain management. Br J Surg. 2020 Jan;107(2):e70-e80. doi: 10.1002/bjs.11477. PMID 31903595